CLINICAL TRIAL: NCT02161042
Title: The Effect of Blood Transfusion on Endothelial Function
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Shahar Lavi, Interventional Cardiologist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 100344
Record Dates: First submitted 2014-06-06; First posted 2014-06-11 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: MDS; Anemia
Keywords: Blood transfusion; Storage Lesion; Endothelial dysfunction; Nitric Oxide
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- fresh blood Transfusion
- Old blood transfusion

SUMMARY:
Blood transfusion is often used to treat patients with Anemia. The period of storage of blood products prior to use for transfusion may vary. Prolonged storage of blood products may result in changing their biochemistry.

This study aims to look into whether the transfusion of "old" blood, which is stored for more than 7 days, as compared to the transfusion of "Fresh" blood, which is stored for less than 7 days, will affect endothelial function.

DETAILED DESCRIPTION:
Endothelial function assessed pre and post transfusion. The EndoPAT uses a unique bio-sensors that are placed on the fingertips to measure pressure. The test takes about 20-25 minutes. During the procedure the participant will have biosensors placed on the index finger of each hand. The nondominant arm will have a blood pressure cuff applied with sufficient pressure for five minutes. At the end of the test the device will provide a reading that assesses the level of endothelial function/dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Age is > 18 years
* Need recurrent blood transfusion

Exclusion Criteria:

* Latex Allergy
* Life expectancy is less than 6 months
* History or evidence of drug or alcohol abuse in the last 12 months
* Any medical condition that will place the participant at a higher risk if they participate in the study

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who come to IV therapy or Oncology day Unit requiring a blood transfusion
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-08; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Endothelial function | Change in endothelial function compared to baseline. Test is done 15 minutes prior to transfusion and 30 minutes post blood transfusion. The test is repeated when patient received another blood transfusion. The results of the change are compared.
  The function of the blood vessels will be assessed with the EndoPAT device. This test is done 15 minutes prior to the transfusion and again 30 minutes post the transfusion. Patients that will receive both fresh and old blood will be included.

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Background] Donadee C, Raat NJ, Kanias T, Tejero J, Lee JS, Kelley EE, Zhao X, Liu C, Reynolds H, Azarov I, Frizzell S, Meyer EM, Donnenberg AD, Qu L, Triulzi D, Kim-Shapiro DB, Gladwin MT. Nitric oxide scavenging by red blood cell microparticles and cell-free hemoglobin as a mechanism for the red cell storage lesion. Circulation. 2011 Jul 26;124(4):465-76. doi: 10.1161/CIRCULATIONAHA.110.008698. Epub 2011 Jul 11. PMID 21747051
- [Background] Kim-Shapiro DB, Lee J, Gladwin MT. Storage lesion: role of red blood cell breakdown. Transfusion. 2011 Apr;51(4):844-51. doi: 10.1111/j.1537-2995.2011.03100.x. PMID 21496045
- [Background] Chin-Yee I, Arya N, d'Almeida MS. The red cell storage lesion and its implication for transfusion. Transfus Sci. 1997 Sep;18(3):447-58. doi: 10.1016/S0955-3886(97)00043-X. PMID 10175158